CLINICAL TRIAL: NCT01365962
Title: A Study to Assess and Quantify Surface Insulin-like Growth Factor I Receptor (IGF-IR) in Rhabdomyosarcoma (RMS) Tumor Tissue
Brief Title: Biomarker in Tumor Tissue Samples From Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST11B4; COG-ARST11B4 (Other: Children's Oncology Group); NCI-2011-02858 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST11B4 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; embryonal childhood rhabdomyosarcoma; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gene Expression Profiling; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in tumor tissue samples from patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine and quantify the degree of surface insulin-like growth factor I receptor (IGF-IR) expression in rhabdomyosarcoma (RMS) tumor tissue.
* To assess the feasibility and validity of a mass spectrometry assay for IGF-IR expression on paraffin-embedded tumor tissue.

OUTLINE: Paraffin-embedded tumor tissue slides are analyzed for insulin-like growth factor I receptor (IGF-1R) expression by mass spectrometry and correlated with the results obtained by IHC assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of rhabdomyosarcoma

  * Alveolar or embryonal rhabdomyosarcoma
* Available samples from the Cooperative Human Tissue Network (CHTN) bank

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of rhabdomyosarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Degree of surface IGF-IR expression in RMS tumor tissue
Feasibility and validity of a mass spectrometry assay for IGF-IR expression on paraffin-embedded tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Suman Malempati, MD, Principal Investigator — Doernbecher Children's Hospital at Oregon Health and Science University